CLINICAL TRIAL: NCT05149417
Title: Effect of Telemedecine on Post-trauma Pain Medication Adherence After Discharge From Emergency Departement
Brief Title: Effect of Telemedecine on Post -Trauma Pain Medication Adherence .
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, chief of the Emergency departement in CHU fattouma Bourguiba Monastir , PhD, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Telemedecine /Adherence
Record Dates: First submitted 2021-11-18; First posted 2021-12-08 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Post-traumatic Pain
Keywords: Telemedecine; Adherence; post- traumatic pain

STUDY DESIGN:
Intervention Model Description: Included patients were randomized to one of the 3 groups:
  1. Usual care (control) group Patients enrolled in this group were discharged and they didn't undergo any intervention within the treatment period.
  2. SMS group Or short message service (SMS) group: patients received SMS at day 2 every day to remind them to take their treatment .
  3. Telemonitoring group:
  Patients received a phone call on day 2 and day 4 to evaluate the adherence , to detect any problem that can affect the adherence to the treatment and modify the analgesic protocol treatment if needed according to an algorithm:
  At each call (day 2 and day 4), the VAS was assessed. If VAS ≥ 3 we looked for a medication discontinuation, inadequate dose or change of the prescribed treatment and the patient was instructed to take action accordingly . If the problem is related to side effects, the analgesic treatment was changed or associated to another analgesic
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard group (Placebo Comparator): Patients enrolled in this group were discharged and they didn't undergo any intervention within the treatment period.
  Interventions: Other: telemonitoring
- SMS group (Active Comparator): patients received SMS at day 2 , day 4 and day 7 after emergency departement discharge to remind them to take their treatment .
  Interventions: Other: SMS reminding
- telemonitoring group (Active Comparator): Patients received a phone call on day 2 and day 4 to evaluate the adherence , to detect any problem that can affect the adherence to the treatment and modify the analgesic protocol treatment if needed.
  Interventions: Other: telemonitoring

INTERVENTIONS:
Other: SMS reminding — patients received SMS at day 2 , day 4 and day 7 after emergency departement discharge to remind them to take their treatment .
  Arms: SMS group
Other: telemonitoring — Patients received a phone call on day 2 and day 4 to evaluate the adherence , to detect any problem that can affect the adherence to the treatment and modify the analgesic protocol treatment if needed.
  Arms: Standard group; telemonitoring group

SUMMARY:
The impact of telemonitoring on patients' adherence to post trauma pain treatment , their satisfaction and pain relief after discharge from the ED.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized trial . Participants are recruited from the emergency departement of Fattouma Bourguiba Monastir.

This study is a seven day three-arm parallel group trial . Participants inculded are aged more than 16 years old who presented to the ED for minor trauma and discharged with analgesic treatment. They are randomized to one of two trial TM intervention groups (SMS and TM) or usual care group (control) in a 1 :1 :1 allocation ratio.

For all inculded patients, demographic characteristics were collected as well as clinical examination findings. The interventional care provided at the ED was mentioned. At ED discharge the pain Visual Analogue Scale (VAS) was evaluated and the analgesic treatment prescribed was noted.

ELIGIBILITY:
Inclusion Criteria:

* Age >16 years old with minor trauma and discharged with an analgesic treatment.
* Included patients should have regular access to a mobile phone ,were able to interact with SMS or could do so with help of a relative.
* Patients who accepted to participate to the study.
* No contraindication to analgesic medication

Exclusion Criteria:

* Swallowing disorder or inability to swallow.
* Unsuitable for follow-up.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1350 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2022-05-21 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Visual analog scale after 7 days of follow-up | at seven day after ED discharge .
  Patient's adherence to analgesics treatment which was assessed by calling patients or by sending SMS in day 2, day 4,and day 7 in SMS group and the telemonitoring group respectively.

SECONDARY OUTCOMES:
Likert scale | at seven day post ED discharge .
  Patients' satisfaction which was assessed through likert scale. minimum=1(strongly disagree) , maximum=5 (strongly agree)

CONTACTS AND LOCATIONS:
Locations (2):
- Tunisia (2):
  - Fattouma Bourguiba Monastir University Hospital Center, Monastir
  - Fattouma Bourguiba University Hospital of Monastir, Monastir

IPD SHARING:
Plan to Share IPD: Undecided